CLINICAL TRIAL: NCT01945190
Title: Acupuncture for Inflammatory Pain and Central Sensitization - A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Nicholas Phillips, MD Candidate, University of Vermont
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 14-079; 28064 (Other: Stanford University)
Record Dates: First submitted 2013-09-04; First posted 2013-09-18 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-10

CONDITIONS: Pain; Inflammation
MeSH Terms: conditions — Pain; Inflammation | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- True before sham electroacupuncture (Experimental): Crossover design, individuals randomized to receive either true or sham acupuncture in first study day, and on the second study day whichever intervention was not administered on the first study day.
  Interventions: Device: Electroacupuncture
- Sham before true electroacupuncture (Experimental): Crossover design, individuals randomized to receive either true or sham acupuncture in first study day, and on the second study day whichever intervention was not administered on the first study day.
  Interventions: Device: Electroacupuncture

INTERVENTIONS:
Device: Electroacupuncture

SUMMARY:
Acupuncture is used extensively by patients worldwide for a variety of illnesses. While research is beginning to show effectiveness in clinical pain, the mechanisms underlying how these effects are evoked are poorly understood. Experimental models in healthy human volunteers can more closely control the variables of acupuncture needling and begin to separate out the relative contribution of specific components of needling and needle stimulation. By examining acupuncture's effects on experimental inflammatory models with well-characterized physiologic mechanisms, hypotheses can begin to be generated regarding how acupuncture produces its clinical effects. We propose to establish a model which could be used as a template to examine the individual components contributing to acupuncture's clinical effects on inflammation and pain. We hypothesize that acupuncture will have analgesic and anti-inflammatory effects on a ultraviolet B induced cutaneous lesion as well as a model of heat pain testing which activates central sensitization.

Twenty healthy human volunteers will participate in a crossover study with active acupuncture and sham acupuncture interventions. They will be tested for their minimal erythemal dose (MED) to ultraviolet B exposure. An experimental lesion at 3x MED will be administered on the lower leg. Background information will be collected which could affect individuals' sensitivity to pain such as anxiety and depression, as well as their expectations regarding acupuncture treatment.

The following day they will return for the first experimental day. A measurement with Laser Doppler will quantify the inflammation in the ultraviolet B lesion. Heat pain testing will be performed using a computer controlled thermode both on and off the ultraviolet B lesion. On-lesion testing will be for heat pain threshold. Off-lesion testing will examine temporal summation of heat pain.

Next, a licensed acupuncturist will perform either true electroacupuncture or sham electroacupuncture in the region adjacent to the ultraviolet B lesion. Participants are blinded to the intervention, as is the examiner collecting data. Afterwards, Laser Doppler and heat pain testing will be repeated. The difference between pre-acupuncture and post-acupuncture measurements will represent the acupuncture -induced analgesic and anti-inflammatory effects.

Participants will return for another ultraviolet B exposure adjacent to the first, and will receive whichever sham or true acupuncture intervention was not performed on the first study day.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-70

Exclusion Criteria:

* Clinically relevant systemic diseases such as psychiatric, neurological, and dermatological conditions interfering with the collection and interpretation of study data
* Chronic or recent use of medication potentially interfering with pain processing (except oral contraceptives)
* Intake of analgesics within the two days prior to study
* Participation in other research studies within the previous 30 days
* Having previously received acupuncture treatments

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Erythema as measured by Laser Doppler | within one day
  Participants are studied in two separate sessions each contained within one day, and each lasting approximately 3 hours. Participants' pre-acupuncture treatment data are compared to post-acupuncture data to assess effect of acupuncture
Heat pain threshold (deg C) | within one day
  Participants are studied in two separate sessions each contained within one day, and each lasting approximately 3 hours. Participants' pre-acupuncture treatment data are compared to post-acupuncture data to assess effect of acupuncture
Analgesia to temporal summation of heat pain | within one day
  Temporal summation of pain is an increased magnitude of response to repetitive stimulus administration. Participants are studied in two separate sessions each contained within one day, and each lasting approximately 3 hours. Participants' pre-acupuncture treatment data are compared to post-acupuncture data to assess effect of acupuncture

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Phillips, BS, BA, MTOM, Principal Investigator — University of Vermont; Helene Langevin, MD, Study Director — University of Vermont
Locations (1):
- Stanford University, Stanford, California, United States